CLINICAL TRIAL: NCT04225000
Title: Effects of Tibiofemoral Mobilization in Patients of Patellofemoral Pain Syndrome
Brief Title: Tibiofemoral Mobilization in Patellofemoral Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00567 Ishrat
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: Tibiofemoral Mobilization; Kujala Anterior Knee Pain Scale; Numeric Pain Rating Scale; Pressure Pain Threshold
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized Control Trail
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Active Comparator): Hip & Knee Exercises
  Interventions: Other: Exercise Group
- Mobilization Group (Experimental): Tibiofemoral joint anterior-posterior mobilization combined Hip & Knee Exercises
  Interventions: Other: Mobilization Group

INTERVENTIONS:
Other: Exercise Group — Control group included 6 different exercises to treat participants having PFPS. These exercises included Semi squat with hip adduction and internal rotation, Quads isometrics, Straight Leg Raise (SLR) Hamstring Stretch, Terminal knee extension with elastic band , Adductor squeeze in crook lying (squeeze the ball), Hip abduction in standing with elastic band. These all exercises were advised to perform 3 x 15 Repetitions with 10 sec hold. This exercise protocol was for 4 weeks and 3 sessions per week.
  Arms: Exercise Group
Other: Mobilization Group — Experimental group included Anterior-Posterior (AP) tibiofemoral joint mobilization and all 6 exercises suggested controlled group for treating participants having PFPS; 3 sessions of mobilizations per week and total 4 weeks.
  These exercises included Semi squat with hip adduction and internal rotation, Quads isometrics, Straight Leg Raise (SLR) Hamstring Stretch, Terminal knee extension with elastic band , Adductor squeeze in crook lying (squeeze the ball), Hip abduction in standing with elastic band. Theses all exercises were advised to perform 3 x 15 Repetitions with 10 sec hold. This protocol was for 4 weeks and 3 sessions per week.
  Arms: Mobilization Group

SUMMARY:
The aim of this research was to determine the effects of tibiofemoral joint mobilization in patients of patellofemoral pain syndrome. Tibiofemoral joint mobilization effects on pain and Range of Motion (ROM) in knee joint. A randomized controlled trial was done at Lady Reading Hospital Peshawar and Hayatabad Medical Complex Peshawar. The sample size was 52. The Participants were divided into two groups, 26 participants in experimental group and 26 in control group. The study duration was 4 months. Sampling technique applied was purposive non probability sampling technique. Only 25 to 35 years participants with patellofemoral pain syndrome were included. Tools used in this study were Numerical pain rating scale (NPRS), Kujala Score Questionnaire, Goniometer and Algometer.

DETAILED DESCRIPTION:
Patellofemoral pain syndrome (PFPS) is the most common overuse injury characterized by anterior and peripatellar knee pain, associated with physical activities in Active Daily Living (ADL) such as climbing stairs, squatting, jumping, and running and by sitting with the knees flexed for prolonged periods of time. It mainly affects young women without any structural changes such as increased Q-angle or significant pathological changes in articular cartilage. It mainly affects young women without any structural changes such as increased Q-angle or significant pathological changes in articular cartilage. Patellofemoral pain has prevalence of 23% in adults and 29% in adolescents annually in general population. Its incidence is higher in women as compare to men and is located at 22/1000 person per year. It accounts for 25-40% of all knee complaints in sports medicine. The prevalence of this problem is high because it can occur in patients with a wide range of physical activity levels.

The main symptom of PFPS is anterior knee pain or pain around and behind patella during patellofemoral joint loading activities. The pathophysiology of PFPS is multifactorial. External factors; change in training intensity and frequency, training surfaces and inappropriate shoe wear, while intrinsic factors includes muscle and soft tissue imbalance and malalignment of lower extremity and poor biomechanics of foot. In PFPS patients' dynamic valgus and patellar maltracking is common. Decrease strength of hip abductors, abnormal rear foot eversion can cause dynamic valgus. Further other muscles imbalance is also associated with PFPS i.e. vastus medialis, vastus lateralis, quadriceps, hamstring and iliotibial tract.

Correction of biomechanical imbalance and decreased anterior knee pain as therapeutic exercise has already been shown to be effective in the treatment of PFPS for pain and function. Conservative treatment involves a multimodal physiotherapy approach including patient education, activity modification, neuromuscular electric stimulation on quadriceps, therapeutic ultrasound, biofeedback, exercises for enhancing the activity of Vastus Medialis Obliquus (VMO) muscle, lower extremity-strengthening exercises, and proximal stabilization, stretching exercises on tight structures, bracings, foot orthoses, patellar mobilization and taping techniques. Patellofemoral pain syndrome is treated through conservative methods from long period of time but

tibiofemoral mobilization is not practiced very much while standard mobilization is patellar mobilization, it can be painful to mobilize patella. So the goal of this study is determine the effect of reciprocal joint mobilization i.e. tibiofemoral joint mobilization in patellofemoral joint pain syndrome and enhance the awareness of this in practice.

Literature review A systematic and evidence based search of relevant literature was performed by utilizing PubMed and Google Scholar as search engines. Search term for the initial literature review was patellofemoral Pain Syndrome, Tibiofemoral mobilization, prevalence of patellofemoral pain syndrome, causes of PFPS, pathophysiology of PFPS, treatment option for PFPS, conservative treatment of PFPS, short term effect of Tibiofemoral mobilization, exercise protocol of PFPS. The search was limited to papers in English preferably published since 2010 with full text available. Different studies were available regarding PFPS but limited data were available regarding tibiofemoral mobilization in PFPS.

A consensus statement (2018) on exercise therapy and physical interventions and mentioned that it is recommended that exercise targeting the hip and knee is a key component of management for all patients with patellofemoral pain, particularly when used in combination.

A consensus statement (2016) from the 4th International Patellofemoral Pain Research Retreat, that exercises are best to treat PFPS in short medium and long term goal and also mentioned that instead of only giving exercises of knee alone if combined hip and knee exercises would be given to patient it will show great effect.

The short-term effects of Movement With Mobilization (MWM) and Kinesio Tapping practices performed in addition to the exercises proved to be similar to one another.

The tibiofemoral joint manipulation with exercises for home plane give a successful results in treating patellofemoral pain syndrome.

A systemic review mentioned that the different combinations of Manual Therapy (MT) and physical therapy analyzed in this review suggest that giving more emphasis to proximal stabilization and full kinetic chain treatments in PFPS will help better alleviation of symptoms.

Another study concluded that interventions directed at the lumbopelvic region did not have immediate effects on quadriceps force output or activation. Muscle fatigue might have contributed to decreased force output and activation over 1 hour of testing.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of anterior knee pain for at least 1 month.
* Anterior or retropatellar knee pain on at least 2 of the following activities: prolonged sitting, climbing stairs, squatting, running, kneeling, and hopping/jumping.
* Presence of 2 of the following clinical criteria on assessment: pain during apprehension test, pain during the patellar compression test, and crepitation during the compression test.

Exclusion Criteria:

* Previous knee surgery or arthritis
* History of patellar dislocation or subluxation, malalignment, or ligament laxity
* Spinal referred pain
* History of other abnormalities such as leg length inequalities (.2 cm)
* Medication as a part of the treatment
* Previous physical therapy or acupuncture treatment for the knee within the previous 30 days.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2019-11-08 (Actual); Study Completion 2020-01-07 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 4th week
  Changes from base Line Numeric Pain Rating Scale is a scale for pain starting from 0-10. where 0 indicate no pain and 10 indicate severe pain
Range Of Motion of Knee Joint (Flexion) | 4th week
  Changes from the Baseline ROM range of Motion of knee joint flexion was taken with the Help of Goniometer
Range Of Motion of Knee Joint (Extension) | 4th week
  Changes from the Baseline ROM range of Motion of knee joint extension was taken with the Help of Goniometer
Pressure Pain Threshold (PPT) | 4th week
  Changes from the Baseline Pressure Pain Threshold (PPT) were taken with the help of Algometer

SECONDARY OUTCOMES:
Kujala Anterior Knee Pain Scale | 4th week
  Changes from the Baseline Kujala Score for Functional activities. Score starting from 0-100.The zero score indicates the greater limitation of knee function whereas the score 100 indicates the ability to perform most knee function.Score were categorized into different functional activities i.e. Limp, weight bearing, pain, stairs climbing, walking, running, jumping, prolonged sitting with knee bent, swelling, atrophy of thigh, loss of knee bend,feeling of instability in knee cap, squatting

CONTACTS AND LOCATIONS:
Overall Officials: Saira Waqqar, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Lady Reading Hospital, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Collins NJ, Barton CJ, van Middelkoop M, Callaghan MJ, Rathleff MS, Vicenzino BT, Davis IS, Powers CM, Macri EM, Hart HF, de Oliveira Silva D, Crossley KM. 2018 Consensus statement on exercise therapy and physical interventions (orthoses, taping and manual therapy) to treat patellofemoral pain: recommendations from the 5th International Patellofemoral Pain Research Retreat, Gold Coast, Australia, 2017. Br J Sports Med. 2018 Sep;52(18):1170-1178. doi: 10.1136/bjsports-2018-099397. Epub 2018 Jun 20. PMID 29925502
- [Background] Briani RV, Pazzinatto MF, De Oliveira Silva D, Azevedo FM. Different pain responses to distinct levels of physical activity in women with patellofemoral pain. Braz J Phys Ther. 2017 Mar-Apr;21(2):138-143. doi: 10.1016/j.bjpt.2017.03.009. Epub 2017 Mar 17. PMID 28460712
- [Background] Crossley KM, van Middelkoop M, Callaghan MJ, Collins NJ, Rathleff MS, Barton CJ. 2016 Patellofemoral pain consensus statement from the 4th International Patellofemoral Pain Research Retreat, Manchester. Part 2: recommended physical interventions (exercise, taping, bracing, foot orthoses and combined interventions). Br J Sports Med. 2016 Jul;50(14):844-52. doi: 10.1136/bjsports-2016-096268. Epub 2016 May 31. No abstract available. PMID 27247098
- [Background] Santos TR, Oliveira BA, Ocarino JM, Holt KG, Fonseca ST. Effectiveness of hip muscle strengthening in patellofemoral pain syndrome patients: a systematic review. Braz J Phys Ther. 2015 May-Jun;19(3):167-76. doi: 10.1590/bjpt-rbf.2014.0089. Epub 2015 May 29. PMID 26039034
- [Background] Demirci S, Kinikli GI, Callaghan MJ, Tunay VB. Comparison of short-term effects of mobilization with movement and Kinesiotaping on pain, function and balance in patellofemoral pain. Acta Orthop Traumatol Turc. 2017 Dec;51(6):442-447. doi: 10.1016/j.aott.2017.09.005. Epub 2017 Oct 17. PMID 29054803
- [Background] Lantz JM, Emerson-Kavchak AJ, Mischke JJ, Courtney CA. TIBIOFEMORAL JOINT MOBILIZATION IN THE SUCCESSFUL MANAGEMENT OF PATELLOFEMORAL PAIN SYNDROME: A CASE REPORT. Int J Sports Phys Ther. 2016 Jun;11(3):450-61. PMID 27274430
- [Derived] Fatimah I, Waqqar S. Effects of tibiofemoral mobilization in patients of Patellofemoral pain syndrome. J Pak Med Assoc. 2021 Nov;71(11):2506-2510. doi: 10.47391/JPMA.04-585. PMID 34783726